CLINICAL TRIAL: NCT02830607
Title: Using Wearable Monitoring Devices for Assessing Efficacy of Epidural Steroid Injection in Patients With Low Back Pain
Brief Title: Wearable Devices to Monitor Efficacy of Epidural Steroid Injection in Patients With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Wiam Welly, Anesthesiology resident, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SHEBA-16-3206-HB-CTIL
Record Dates: First submitted 2016-06-18; First posted 2016-07-13 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Xiaomi Mi Band (Experimental): participants will wear Xiaomi Mi Band .the device measures their daily steps number before and after epidural steroid injection for treatment of low back pain.
  Interventions: Device: Xiaomi Mi Band

INTERVENTIONS:
Device: Xiaomi Mi Band — participants will wear Xiaomi Mi Band as assessment tool for recovery after epidural steroid injection for treatment of low back pain

SUMMARY:
Low back pain (Lower Back Pain ) is extremely common , affecting more than 80 % of the general population in the modern world , one is considered the most common cause of disability in people under the age of 45. Lower back pain represents a social problem and substantial economies in Western countries , also considered a first cause for orthopedic consultation. In recent decades , a number of methods developed for assessing the functional status of patients with low back pain , and over twenty -five generic methods available today for use in pain clinics , orthopedic clinics and in clinical trials A large part of the measures used to monitor the response of patients to treatment of low back pain based on self-report questionnaires ,on patients' pain intensity , quality of life measures , and functional status In recent years a number of wearable monitoring devices designed to help people assess the progress of sports activity , by measuring steps , pulse , and quality of sleep , in this study we will use these measures to assess treatment efficacy after steroid injection to the epidural space in patients with low back pain . And compare the results to those taken from subjective self-report questionnaires .

DETAILED DESCRIPTION:
Low back pain (Lower Back Pain) is extremely common, affecting more than 80% of the general population in the modern world, one is considered the most common cause of disability in people under the age of 45. 2 Lower back pain represents a social problem and substantial economies in Western countries, such as also considered a first cause orthopedic advice ahead. 3 Over the past decades, developed a number of methods for assessing the functional status of patients with low back pain, 4-7 and over twenty-five generic methods available today for use in pain clinics, orthopedic clinics and in clinical trials. 8 A large part of the measures used to monitor the response of patients to treat low back pain based on self-report questionnaires on patients' pain intensity, quality of life measures, and functional status.measures which relate to such measures - reduction of pain, reduction in the consumption of medication relieve pain, improved mood, improved daily function, improved sleep patterns, back in daily life and work, a reduction in the consumption of health system resources, and reduction in disability benefits, sick leave, early retirement, and more. The existence of multiple assessment tools of this type suggests that there is no a single tool valid and reliable for assessing the severity of low back pain and its response to treatment. In addition, there is a problematic depending on the patient's self-report is subjective and often biased because of the possibility of secondary gain illness.

In recent years there has been great progress in the use of technologies of wearable monitoring both by the general population as part of the tracking of daily living and sports, as well as in a clinical setting. The use of cheap and simple devices give the user information about the number of steps performed during the day measuring heart rate and sleep quality .

In the present work the investigators will make use of wearable and affordable device that measures a number of steps and sleep quality monitoring recovery after epidural steroid injection for patients with low back pain. The indices will be accepted through this monitoring will be compared with subjective reports of participants and physician's assessment about the success of the treatment. investigators Will use the wearable monitoring type Xiaomi Mi Band for measuring steps and sleep quality the device was chosen because it is cheap, easy to use, has long battery life (two weeks between charges), and the participants can continue to wear it every hour of the day and while bathing. as a measure of subjective filled questionnaire by the participants,the investigators selected the Oswestry Disability Index (ODI) . This questionnaire addresses aspects of wider life of the patient and is composed of 10 sections: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, socializing, travel and employment.Each section includes values from 0 to 5 , with higher values representing higher functional limitation . The final score is obtained using a standard scoring .

ELIGIBILITY:
Inclusion Criteria:

* After Ethics Committee approval and consent to participate in research. self- aware 40 patients aged 18-60 Hebrew, speakers who come for the first time to a pain clinic for the treatment with epidural steroid injection due to low back pain and express their consent to participate in the study

Exclusion Criteria:

* the study will not include patients who received steroid injection to the epidural space as part of previous treatment, the study will not include morbid obese patients B.M.I over 30, patients with symptomatic coronary artery disease, patients with known osteoarthritis that or any orthopedic disease that limit their walking capacity, C.O.P.D patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-21 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
number of steps . | from the day of making the decision for treatment until four weeks after treatment.
  the investigators will be using the xiaomi mi band to measure the number of steps the participants make daily. from the day of making the decision for treatment (steroid injection for epidural space) until four weeks after treatment. this measures will be compared to the score taken from Oswestry disability index (ODI) Before treatment and on day 3,7,14 and 28 after treatment. Evaluating the treatment response by the treating pain physician using a scale from zero to ten, where (zero no response an 10 great response).

CONTACTS AND LOCATIONS:
Overall Officials: Haim Berkenstadt, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li RT, Kling SR, Salata MJ, Cupp SA, Sheehan J, Voos JE. Wearable Performance Devices in Sports Medicine. Sports Health. 2016 Jan-Feb;8(1):74-8. doi: 10.1177/1941738115616917. Epub 2015 Nov 11. PMID 26733594
- [Background] Knowles LM, Skeath P, Jia M, Najafi B, Thayer J, Sternberg EM. New and Future Directions in Integrative Medicine Research Methods with a Focus on Aging Populations: A Review. Gerontology. 2016;62(4):467-76. doi: 10.1159/000441494. Epub 2015 Nov 7. PMID 26545038
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Longo UG, Loppini M, Denaro L, Maffulli N, Denaro V. Rating scales for low back pain. Br Med Bull. 2010;94:81-144. doi: 10.1093/bmb/ldp052. Epub 2010 Jan 10. PMID 20064820
- [Background] Grotle M, Brox JI, Vollestad NK. Functional status and disability questionnaires: what do they assess? A systematic review of back-specific outcome questionnaires. Spine (Phila Pa 1976). 2005 Jan 1;30(1):130-40. PMID 15626993
- [Background] Luo X, Pietrobon R, Sun SX, Liu GG, Hey L. Estimates and patterns of direct health care expenditures among individuals with back pain in the United States. Spine (Phila Pa 1976). 2004 Jan 1;29(1):79-86. doi: 10.1097/01.BRS.0000105527.13866.0F. PMID 14699281